CLINICAL TRIAL: NCT02857322
Title: Effectiveness Accompaniment Perioperative Patients With Psychiatric Illness on the Lives Perioperative
Acronym: VEPSY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014-48
Record Dates: First submitted 2016-07-29; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subjects with documented psychiatric pathology (Other)
  Interventions: Other: Accompanying patient's specific perioperative

INTERVENTIONS:
Other: Accompanying patient's specific perioperative

SUMMARY:
The experimental strategy is to develop a specific device about the anesthetic and surgical acts for a subject with a documented psychiatric condition and to benefit from surgery. This device is based on 3 stages: pre-operative phase, Phase perioperative and postoperative phase. A nurse anesthetist will come into contact with the subject the day before surgery. This contact will be concomitant with the pre-anesthesia visit. She explained about the general organization of the arrival in the operating room. The interview will be a minimum of 15 minutes and beyond if necessary. This will be accompanying this the next day in the operating room in order to optimize its hospitality and installing the block, guide the subject through all the steps before falling asleep. Finally, even accompanying will be present upon awakening the subject in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* adult subject;
* Subject with chronic mental illness defined by ICD-10 classification [ICD-10, 1992], corresponding to psychoses say no emotional or affective psychoses say;
* Subject to which mental pathology is evolving for more than 6 months;
* Topic targeted for elective surgery;
* Topic judged capable of performing a self-administered questionnaire;

Exclusion Criteria:

* minor, pregnant or nursing women, about not being affiliated to the social security scheme, subject under guardianship;
* Subject with a mental illness do not belong to sections of ICD-10 contained in "inclusion criteria";
* Subject to benefit from surgery as part of the emergency;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-01 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
experiences of the perioperative period | second day
  assessment using a self-administered questionnaire called EVAN. This is a standardized questionnaire and validated, whose purpose is to understand the experience of perioperative anesthesia multidimensional way. It contains 28 items describing 6 dimensions (anxiety, discomfort, fear, pain and discomfort, explanations, needs). dimensional scores range from 0 (worst experience) to 100 (best experience).

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France